CLINICAL TRIAL: NCT06968598
Title: Analysis of Early Neurodevelopmental Alterations in Bipolar Disorder Based on Cortical Organoid Models
Acronym: BIPODEV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A02158-39
Record Dates: First submitted 2024-12-19; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Bipolar Disorder (BD); Organoids; Neurodevelopmental Conditions
Keywords: organoid; neurodevelopmental alterations
MeSH Terms: conditions — Bipolar Disorder | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurodevelopmental alteration (Experimental): blood sampling to generate organoids in the ND group
  Interventions: Other: blood sample
- No Neurodevelopmental alteration (Placebo Comparator): blood sampling to generate organoids in the non- ND group
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — blood sample

SUMMARY:
Demonstrate the existence of neurodevelopmental alterations in organoids derived from samples of patients with bipolar disorder (BD) with a neurodevelopmental (ND) component, compared with patients with bipolar disorder (BD) without an ND component.

ELIGIBILITY:
Inclusion Criteria:

* Presence of bipolar disorder according to DSM-5 criteria
* Able to freely give and sign consent
* Affiliated or beneficiary of a health insurance plan
* Previous participants in the NEMO study (2022-A00353-40)

For the "neurodevelopmental bipolar" (ND-BP) group: presence of a neurodevelopmental burden score in the top 5, as assessed in the NEMO project (NCT05674019).

For the "non-neurodevelopmental bipolar" group (TB): presence of a neurodevelopmental load score of 0, or in the lowest 5, as assessed in the NEMO project.

Exclusion Criteria:

* - Presence of a severe symptomatic or unstable physiological or medical condition (including pregnancy)
* History of psychiatric illness (stable or not), schizophrenia or any other pathology likely to interfere with bipolar disorder
* History of severe head trauma (GCS<8 at time of trauma)
* Presence of a neurological disorder affecting central nervous system function
* Presence of moderate to severe substance use disorders (>=4/11 as defined in DSM-5), with the exception of tobacco use disorders.
* The volunteer is under court protection or guardianship
* It proves impossible to give the volunteer informed information, or the volunteer refuses to sign the consent form.
* Insufficient command of the French language to complete evaluations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the existence of neurodevelopmental alterations in organoids derived from samples of patients with bipolar disorder with a neurodevelopmental (ND) component, compared with patients with bipolar disorder without ND component. | Through study completion, an average of 2 year
  Organization of cortical layers in both subgroups

SECONDARY OUTCOMES:
Establish induced pluripotent stem cell (iPSC) lines from cryopreserved PBMCs of the TB-ND subgroup | Through study completion, an average of 2 year
  Pluripotency
Quality of cortical organoids produced from these iPSCs | Through study completion, an average of 2 year
  Viability of organoids
Assessing the reproducibility of the iPSC derivation protocol in cortical organoids | Through study completion, an average of 2 year
  Reproducibility of the cortical organoid differentiation protocol

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Director of the AP-HM

IPD SHARING:
Plan to Share IPD: Undecided